CLINICAL TRIAL: NCT07193576
Title: A Randomized, Open-Label, Two-Period, Two-Crossover Study to Evaluate the Effect of Food on the Pharmacokinetics of Flonoltinib Maleate Tablets in Healthy Subjects Under Fed Conditions
Brief Title: A Pharmacokinetic Study of the Food Effect on Flonoltinib Maleate Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chengdu Zenitar Biomedical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: H-FNTN-PI-FE
Record Dates: First submitted 2025-04-02; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Heathly Subjects
Keywords: Flonoltinib Maleate Tablet; Pharmacokinetic study; Heathly Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A group (Experimental): Subjects received Flonoltinib Maleate: under fast condition → washout → under fed condition
  Interventions: Drug: flunotinib
- B group (Experimental): Subjects received Flonoltinib Maleate: under fed condition → washout → under fast condition
  Interventions: Drug: flunotinib

INTERVENTIONS:
Drug: flunotinib — 100mg

SUMMARY:
A Randomized, Open-Label, Two-Period, Two-Crossover Study to Evaluate the Effect of Food on the Pharmacokinetics of Flonoltinib Maleate Tablets in Healthy Subjects Under Fed Conditions

DETAILED DESCRIPTION:
Primary Study Objective. To evaluate the effect of a high-fat diet on the pharmacokinetics of single-dose oral Flonoltinib Maleate tablets in healthy subjects.

Secondary Study Objectives To evaluate the safety of single-dose oral administration of Flonoltinib Maleate Tablets under Fast or Fed condition in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 45 years old (including 18 and 45 years old), gender is not limited;
2. Male subjects weighing ≥50.0 kg, female subjects ≥45.0 kg, with body mass index (BMI) between 19.0 and 25.0 kg/m2 (including borderline values);
3. Fully understand the content of the trial, the test drug, the trial process, etc, and be able to communicate well with the researcher, willing to comply with the study regulations, participate in the trial voluntarily and sign an Inform consent.

Exclusion Criteria:

1. Those with a history of severe allergies (e.g, angioedema and anaphylaxis), allergies (Screening Consultation/Admission Consultation) Those with a history of severe allergy (e.g, angioedema and anaphylaxis), allergy (e.g, allergy to pollen, two or more medications/foods), or history of food or drug allergy or other metabolic disorders (e.g, asthma, hives, eczematous dermatitis, etc.) judged by the investigator to be clinically significant, or a known allergy to JAK inhibitors or an allergy to excipient components of the test medication;
2. Abnormal and clinically significant results of physical examination, vital signs, 12-lead electrocardiogram, laboratory tests (including routine blood, blood biochemistry, urine routine, blood pregnancy (only for women of childbearing age), infectious disease screening, antinuclear antibody, coagulation function, tuberculosis antibody, chest X-ray, abdominal ultrasound) prior to enrolment;
3. QTcF > 440 ms for males and > 460 ms for females on ECG during the screening period;
4. Those who have undergone major surgical procedures within 3 months prior to screening or plan to undergo surgery during the trial period;
5. Acute illness within 2 weeks prior to screening; clinically significant infection (e.g, upper respiratory tract infection, nasopharyngitis, urinary tract infection, etc.) within 3 months prior to screening; evidence of any infection within 7 days prior to screening; history of herpes simplex infection, or recurrent (>once) herpes zoster or disseminated herpes zoster;
6. History of any clinically serious disease or any disease or condition that, in the opinion of the investigator, may affect the outcome of the trial, including but not limited to a history of circulatory, endocrine, neurological, gastrointestinal, urinary, or haematological, immunological, psychiatric, and metabolic disorders;
7. Dysphagia or any history of gastrointestinal disorders (or gastrointestinal resection, etc.) affecting drug absorption; 8 . Those with irregular bowel movements and habitual constipation or diarrhoea;

9. Those with a history of lipid metabolism defects, such as: familial hyperlipidaemia, lipoid nephropathy, or patients with acute pancreatitis accompanied by hyperlipidaemia; 10. Those with a positive combined urine multi-drug test (including morphine, methamphetamine, ketamine, methylenedioxyamphetamine, tetrahydrocannabinolic acid); 11. Those with a history of previous drug abuse or drug dependence; 12. Anyone who has been vaccinated within 8 weeks prior to screening or who plan to be vaccinated during the course of the study or within 8 weeks of administration of study drug; 13. Anyone who has donated or lost ≥400 mL of blood or received a blood transfusion within 3 months prior to screening; or anyone who has donated blood or blood components within 1 month of the planned end of the trial; 14. Those with special dietary requirements or those who are unable to comply with the uniform dietary and appropriate regulations of the study center; 15. Those who have smoked more than 3 cigarettes/day or equivalent amount of tobacco in the 3 months prior to screening; or who have consumed ≥14 units of alcohol per week (1 unit equals to 17.5mL or 14g of pure alcohol, which is approximately equal to 35mL of 50° white wine or 350mL of 5° beer); or who do not agree to abstain from smoking or drinking alcohol for the duration of the trial; or those who have a positive result from an alcohol breathalyzer test; 16. Any person who has taken any prescription drug, over-the-counter drug, any vitamin product or herbal medicine (JAK inhibitor, immunosuppressant, etc.) within 14 days prior to screening; 17. Those who have combined strong inducers of liver metabolism enzymes (e.g, omeprazole, barbiturates, carbamazepine, amiloride, pallidomycin, aminoglutethimide, phenytoin, grumet, rifampicin, sulfinpyrazone, roxithromycin, etc.) within the 4 weeks (28 days) prior to Screening, or any other history of medication use that in the judgement of the Investigator has the potential to interfere with in vivo pharmacokinetics of the test drug. Anyone who has taken any drug known to cause prolongation of the QT/QTcF interval or a drug with a risk of causing torsades de pointes (TdP) within 4 weeks (28 days) prior to Screening; or drugs with a long half-life; 18. Anyone who consumed any food or drink containing caffeine (e.g. coffee, strong tea, cola, chocolate, etc.) or food containing grapefruit juice that may have an effect on metabolising enzymes or who consumed food or drink containing alcohol within 48 h prior to the administration of the drug; 19. Those who are participating in other clinical trials and have used an investigational drug, vaccine or device within 3 months prior to the first dose; 20. Pregnant or breastfeeding women or women of childbearing age who have had unprotected sex within 14 days prior to screening; 21. The subject or his/her partner is unwilling to use non-pharmacological contraception (e.g, total abstinence, condom, IUD, ligation, etc.) for contraception during the trial period or the subject and/or his/her partner has a pregnancy plan within 3 months of the administration of the study drug; 22. The subject may not be able to complete the study for other reasons or there are other factors that, in the opinion of the investigator, make participation in the trial unsuitable.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-08-04 (Actual); Primary Completion 2024-09-11 (Actual); Study Completion 2024-09-11 (Actual)

PRIMARY OUTCOMES:
Cmax | Day1 and Day11 Within 2hours before administration and 0.5 hours, 1 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12hours, 24hours, 48 hours, 72 hours, 96 hours, 120hours, 144 hours after administration
  maximum concentration
AUC0-t | Day1 and Day11 Within 2 hours before administration and 0.5 hours, 1 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12hours, 24hours, 48 hours, 72 hours, 96 hours, 120hours, 144 hours after administration
  Area under the blood concentration-time curve from 0 o 'clock to the last measurable concentration at collection time t
AUC0-∞ | Day1 and Day11 Within 2 hours before administration and 0.5 hours, 1 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12hours, 24hours, 48 hours, 72 hours, 96 hours, 120hours, 144 hours after administration
  The area under the blood drug concentration-time curve from 0 to infinity time
Tmax | Day1 and Day11 Within 2 hours before administration and 0.5 hours, 1 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12hours, 24hours, 48 hours, 72 hours, 96 hours, 120hours, 144 hours after administration
  time to peak
t1/2 | Day1 and Day11 Within 2 hours before administration and 0.5 hours, 1 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12hours, 24hours, 48 hours, 72 hours, 96 hours, 120hours, 144 hours after administration
  Terminal phase elimination half-life
tlag | Day1 and Day11 Within 2 hours before administration and 0.5 hours, 1 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12hours, 24hours, 48 hours, 72 hours, 96 hours, 120hours, 144 hours after administration
  retardation time
CL/F | Day1 and Day11 Within 2 hours before administration and 0.5 hours, 1 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12hours, 24hours, 48 hours, 72 hours, 96 hours, 120hours, 144 hours after administration
  apparent clearance
Vd/F | Day1 and Day11 Within 2 hours before administration and 0.5 hours, 1 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12hours, 24hours, 48 hours, 72 hours, 96 hours, 120hours, 144 hours after administration
  apparent volume of distribution
λz | Day1 and Day11 Within 2 hours before administration and 0.5 hours, 1 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12hours, 24hours, 48 hours, 72 hours, 96 hours, 120hours, 144 hours after administration
  Terminal elimination rate constant
%AUCex | Day1 and Day11 Within 2 hours before administration and 0.5 hours, 1 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12hours, 24hours, 48 hours, 72 hours, 96 hours, 120hours, 144 hours after administration
  The extrapolation percentage of AUC0--∞

SECONDARY OUTCOMES:
health checkup | Screening period, day 17 or early withdrawal
  General examination
participants with abnormal vital signs | Screening period,Day1to day7 and day11 to day17
  Temperature
participants with abnormal laboratory tests results | Screening period, Day-1 (examination results within 7 days are acceptable), Day17, or early withdrawal
  White blood cell count
participants with abnormal laboratory tests results | Screening period, Day-1 (examination results within 7 days are acceptable), Day17, or early withdrawal
  creatinine
participants with abnormal laboratory tests results | Screening period, Day-1 ,Day 10,Day 17 or early termination
  Blood pregnancy test,Only for women of childbearing age
Urinary albumin creatinine ratio | D-1, D17 or early termination
  Urinary albumin creatinine ratio
ECG QT Interv | Screening period, Day-1 ,Day1, Day10, Day11, Day17 or early termination
  12-lead electrocardiogram
participants with abnormal vital signs | Screening period,Day1to day7 and day11 to day17
  blood pressure
participants with abnormal laboratory tests results | Screening period, Day-1 (examination results within 7 days are acceptable), Day17, or early withdrawal
  neutrophil count
participants with abnormal laboratory tests results | Screening period, Day-1 (examination results within 7 days are acceptable), Day17, or early withdrawal
  hemoglobin
participants with abnormal laboratory tests results | Screening period, Day-1 (examination results within 7 days are acceptable), Day17, or early withdrawal
  platelet coun
participants with abnormal laboratory tests results | Screening period, Day-1 (examination results within 7 days are acceptable), Day17, or early withdrawal
  red blood cell count
participants with abnormal laboratory tests results | Screening period, D-1 (examination results within 7 days are acceptable), Day17, or early withdrawal
  alanine aminotransferase
participants with abnormal laboratory tests results | Screening period, D-1 (examination results within 7 days are acceptable), Day17, or early withdrawal
  aspartate aminotransferase
participants with abnormal laboratory tests results | Screening period, Day-1 (examination results within 7 days are acceptable), Day17, or early withdrawal
  total bilirubin
participants with abnormal laboratory tests results | Screening period, Day-1 (examination results within 7 days are acceptable), Day17, or early withdrawal
  direct bilirubin
participants with abnormal laboratory tests results | Screening period, Day-1 (examination results within 7 days are acceptable), Day17, or early withdrawal
  γ-glutamyl transpeptidase
participants with abnormal laboratory tests results | Screening period, Day-1 (examination results within 7 days are acceptable), Day17, or early withdrawal
  Alkaline phosphatase
participants with abnormal laboratory tests results | Screening period, Day-1 (examination results within 7 days are acceptable), Day17, or early withdrawal
  triglycerides
participants with abnormal laboratory tests results | Screening period, Day-1 (examination results within 7 days are acceptable), Day17, or early withdrawal
  total cholesterol
adverse event | From date of randomization until the date of completion of data collection, assessed up to 17 days or early termination
  Adverse events, serious adverse events, suspected and unexpected serious adverse reactions (SUSAR), priority adverse reactions, incidence of adverse reactions
participants with abnormal urinalysis | Screening period, Day-1 , Day17, or early withdrawal
  Acidity/Alkalinity
participants with abnormal urinalysis | Screening period, Day-1 , Day17, or early withdrawal
  Red Blood Cells
participants with abnormal urinalysis | Screening period, Day-1 , Day17, or early withdrawal
  White Blood Cells
participants with abnormal urinalysis | Screening period, Day-1 , Day17, or early withdrawal
  Protein
participants with abnormal urinalysis | Screening period, Day-1 , Day17, or early withdrawal
  Glucose

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolan Yong, bachelor, Principal Investigator — Chengdu Xinhua Hospital
Locations (1):
- Chengdu Xinhua Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No